CLINICAL TRIAL: NCT06128304
Title: ACCESS: Accelerating Cervical Cancer Elimination Through the Integration of Screen-and-treat Services
Acronym: ACCESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Nigeria Nsukka (Other)
Responsible Party: Principal Investigator, Gregory Aarons, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: U01CA275118 (NIH)
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: HIV; Cervical Cancer
Keywords: Implementation Science; Cluster randomized trial; Capacity building; Low and middle income countries; Research infrastructure; Exploration Preparation Implementation Sustainment (EPIS); EPIS Framework
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Implementation Strategies (Active Comparator): Core Implementation Strategies
  1. Ongoing consultation
  2. Educational meetings
  3. Strengthen referral system
  4. Prepare patients to be active participants
  Interventions: Other: Core Implementation strategies; Other: Core+ Enhanced Implementation Strategies
- Core+ Enhanced Implementation Strategies (Experimental): Includes all of the Core implementation strategies and adds:
  5. Community engagement using Health Beginning Initiative Model
  6. Smart Cards to facilitate patient engagement
  Interventions: Other: Core+ Enhanced Implementation Strategies

INTERVENTIONS:
Other: Core Implementation strategies — Core Implementation Strategies
  1. Ongoing consultation
  2. Educational meetings
  3. Strengthen referral system
  4. Prepare patients to be active participants
  Arms: Core Implementation Strategies
Other: Core+ Enhanced Implementation Strategies — Includes all of the Core implementation strategies and adds:
  5. Community engagement using Health Beginning Initiative Model
  6. Smart Cards to facilitate patient engagement

SUMMARY:
While there has been a significant increase in the uptake of antiretroviral therapy among women living with HIV (WLHIV) in many low- and-middle income countries (LMICs), the coverage of cervical cancer screening and treatment (CCST) among WLHIV remains low. This study aims to leverage the available infrastructure for HIV care and treatment programs in Nigeria to integrate cervical cancer screening and treatment and conduct a cluster randomized, hybrid type III trial design to assess the comparative effectiveness of a Core set of implementation strategies versus a Core+ (enhanced) set of implementation strategies to implement cervical cancer screening, onsite treatment, referral and referral completion, treatment, and retention in care among WLHIV. The overarching goal is to improve the health and life expectancy of WLHIV with co-occurring cervical cancer.

DETAILED DESCRIPTION:
Nigeria has one of the largest HIV epidemics in the world with 1.8 million people living with HIV infection. With an estimated female population of 102 million and HIV prevalence of 1.6% among adult females, Nigeria has the largest population of women and the 4th largest number of women living with HIV (WLHIV) in Africa. Although access to antiretroviral therapy (ART) among WLHIV in Nigeria has increased over the years, with over 98% of the 960,000 WLHIV on ART, AIDS-related mortality remains high. In 2020, 16,000 WLHIV died from AIDS- related illnesses including cervical cancer. A pilot implementation program in Nigeria demonstrated that leveraging the U.S. President's Emergency Plan for AIDS Relief (PEPFAR) supported HIV programs for the provision of evidence-based cervical cancer screen-and-treat interventions in WLHIV is feasible. The pilot program demonstrated, however, that tailored implementation strategies will be needed to address specific multilevel barriers along the cancer control continuum in order to address adoption, reach, and sustainability that are necessary for successful scale-up. However, in many African countries with a high burden of both HIV and cervical cancer, there is a paucity of evidence-based implementation strategies to inform effective integration of HIV and cervical cancer services delivery. Objectives of this proposal are to: 1) Refine strategies to integrate cervical cancer screening, treatment and management within existing comprehensive HIV treatment programs and determine implementation readiness; 2) Determine the comparative effectiveness of a Core set of implementation strategies versus Core+ enhanced implementation strategies; and 3) assess sustainment of the integration of cervical cancer screening, treatment, and management intervention into HIV programs. The investigators have assembled a strong team from University of California San Diego, the University of Nigeria, Nsukka, and Northeastern University with expertise in implementation science, HIV care and research, and cancer care and research. Our proposal is responsive to the NCI request for applications (RFA) and consistent with the World Health Organization global plan of elimination of cervical cancer by 2030. If effective, the proposed project will result in a set of feasible, culturally adaptable, and sustainable implementation strategies to integrate evidence-based cervical cancer screening and treatment into HIV programs in order to improve the health and life expectancy of WLHIV.

ELIGIBILITY:
Inclusion Criteria:

* Women living with HIV

Exclusion Criteria:

-

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 2436 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Reach | 12 months after enrollment
  Percent of WLHIV who had cervical cancer (CC) screening
Sustainment | 3 months prior to study completion
  Provider Report of Sustainment Scale (PRESS; Moullin et al., 2021). The PRESS has 3-items scored from 0 "not at all" to 4 "to a very great extent" where higher scores indicate better evidence-based practice sustainment.

SECONDARY OUTCOMES:
CCST Effectiveness | 15 months after treatment of pre-invasive cancer
  Percent of WLHIV treated for pre-invasive cancer who had negative post treatment follow-up screen

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Aarons, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- UC San Diego, La Jolla, California, United States
- University of Nigeria, Nsukka, Enugu, Enugu State, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olakunde BO, Itanyi IU, Olawepo JO, Liu L, Bembir C, Idemili-Aronu N, Lasebikan NN, Onyeka TC, Dim CC, Chigbu CO, Ezeanolue EE, Aarons GA. Comparative effectiveness of implementation strategies for Accelerating Cervical Cancer Elimination through the integration of Screen-and-treat Services (ACCESS study): protocol for a cluster randomized hybrid type III trial in Nigeria. Implement Sci. 2024 Mar 11;19(1):25. doi: 10.1186/s13012-024-01349-9. PMID 38468266